CLINICAL TRIAL: NCT05780658
Title: Feasibility of a Purpose in Life Renewal Intervention for Adults With Persistent Symptoms After Concussion
Acronym: PSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Radomski (Other)
Responsible Party: Sponsor-Investigator, Mary Radomski, Senior Scientific Advisor, Allina Health System
Organization: Allina Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006262
Record Dates: First submitted 2023-03-13; First posted 2023-03-22 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Concussion; Syndrome
MeSH Terms: conditions — Brain Concussion; Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compass Course (Experimental): Four groups of up to 12 participants (48 total) will receive the study intervention during Spring and Fall 2022. All participants will complete study questionnaires before and after the sessions.
  Interventions: Behavioral: Compass Course

INTERVENTIONS:
Behavioral: Compass Course — An 8-session group intervention that integrates education, support, self-reflection, and action-expectation to help people reaffirm or reconstruct self-grounded purpose after significant life events/transitions. The 8 sessions extend over 2-3 months, with 7 weekly sessions and the final session 1 month after Session 7. The intervention, called the Compass Course is structured around the 6 dimensions of flourishing (autonomy, self-acceptance, personal growth, relationships, purpose in life, external mastery), the goal of which is to help people enact behaviors that move them forward in reframing a sense of self and reaffirming or reconstructing a sense of purpose in their daily lives.

SUMMARY:
A group of clinicians and researchers developed an 8-session group intervention that integrates education, support, self-reflection, and action-expectation to help people reaffirm or reconstruct self-grounded purpose after significant life events/transitions. The 8 sessions extend over 2-3 months, with 7 weekly sessions and the final session 1 month after Session 7. The intervention, called the Compass Course is structured around the 6 dimensions of flourishing (autonomy, self-acceptance, personal growth, relationships, purpose in life, external mastery), the goal of which is to help people enact behaviors that move them forward in reframing a sense of self and reaffirming or reconstructing a sense of purpose in their daily lives. Participating in this research will involve an introduction session, where informed consent will be obtained, followed by the 8-session intervention for 9 sessions in total.

A team composed of researchers from Courage Kenny Rehabilitation Institute (CKRI) propose to recruit a convenience sample of individuals who were hospitalized with COVID-19 to evaluate the efficacy of administering the Compass Course to a novel population, to improve psychological well-being, engagement in everyday activities, and purpose in life.

A focus group will be scheduled 2 months after the completion of the Compass Course. This session is composed of brief questionnaires and designed to obtain post-course data to help evaluate the Compass Course intervention.

DETAILED DESCRIPTION:
Aim #1: To evaluate the acceptability of the CC intervention (purpose renewal intervention) delivered via HIPAA-compliant Zoom to adults with PSC who report lacking a sense of direction in life. Quantitative measures of acceptability will include number of inquiries to explore study participation; participant intervention completion rate; participant responses to an Experience Survey at posttest. The investigators will also conduct posttest focus groups to assess aspects of the intervention that may need to be modified prior to a larger study.

Aim #2: To determine the extent to which the CC has beneficial effects on psychosocial outcomes (i.e., self-reported purpose in life; functioning; persistent concussion symptoms) for adults with PSC. The investigators will use a one-group, pretest-posttest design collecting pretest, posttest, and 2-month follow-up data. Main outcomes will include self-reported purpose in life (purpose in life subscale of the Scales of Psychological Wellbeing (Ryff & Keyes, 1995) and Meaning in Life Questionnaire (Steger et al., 2006). Secondary outcomes will include engagement in purpose activities (Life Engagement Test [Scheier et al., 2006]) and concussion symptoms (Rivermead Post Concussion Symptoms Questionnaire [King et al., 1995].

Aim #3: To explore the relationship between participants' real-time responses to purpose prompts delivered via a smartphone app and intervention adherence and outcomes. The investigators will employ mobile ecological momentary assessment to prompt participants to make daily purpose-related choices from the start of the study intervention and evaluate whether participation in these daily prompts is related to primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Response to Purpose Status Question (PSQ) suggests that lack of Purpose Direction
* 18 years or older
* Able to communicate in English
* Evidence of persistent concussion symptoms (concussion symptoms that persist at least 3 months after date of concussion) for concussions occurring in the past 2 years
* Received medical-rehabilitative services for persistent concussion symptoms over the past 12 months based on documentation in EPIC (i.e., ICD9 or ICD10 codes) or clinician referral to the study
* Access to computer or tablet and adequate internet connection to participate in video conference
* Has an email address
* Has a device (computer with webcam, tablet) to use for Zoom access during sessions
* Has access to an internet connection - broadband wired or wireless (3G or 4G/LTE)
* Own a smartphone with one of the following operating system versions:

iOS 9.0 - 9.3, 10.0 - 10.3, 12, 13.3, 13.7, 14.0 - 14.4 or later Android 8.0 - 8.1.0, 9, 10, 11 or later

* Agrees to use personal smartphone to download mEMA application and respond to application notifications (mEMA is described below)
* Agrees to make every effort to attend all group sessions, respond to mEMA notifications many times per week, and to spend 30 minutes each week performing homework

Exclusion Criteria:

* Has significant problems in everyday functioning that would interfere with full participation in the intervention, indicated by a WSAS score above 30 during screening (indicative of severe functional pathology [Mundt et al., 2002]).
* Reports being unable to see, hear, or speak (with or without assistive devices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Purpose in Life | Three months
  Purpose-related subscale of a widely-used self-report questionnaire that was designed to measure 6 theoretically motivated dimensions of psychological well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Courage Kenny Research Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No